CLINICAL TRIAL: NCT01612793
Title: Non-Invasive Vagus Nerve Stimulation With the AlphaCore Device for Management of Bronchoconstriction in Patients Hospitalized With COPD
Brief Title: Vagus Nerve Stimulation for Management of Bronchoconstriction in Patients Hospitalized With COPD Exacerbations
Status: Terminated | Type: Observational
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Other Study IDs: COPD-CA-01
Record Dates: First submitted 2012-05-25; First posted 2012-06-06 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Complete CBC and blood gases will be drawn at different time points to establish the medical condition of the subjects.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AlphaCore device: AlphaCore device group will consist of subjects enrolled into the study with chronic obstructive pulmonary disease and receive an electrical stimulation to the vagus nerve to help open the subjects airways during the subjects stay in the hospital.
  Interventions: Device: AlphaCore Device

INTERVENTIONS:
Device: AlphaCore Device — multiple stimulation treatments per day for duration of hospitalization
  Other Names: Non-invasive vagus nerve stimulation

SUMMARY:
This study will look at the safety, improving symptoms and decreasing the length of stay of patients admitted to the hospital with COPD.

DETAILED DESCRIPTION:
The primary safety measurement for this study is the type, occurrence and severity of adverse events (anticipated and unanticipated), including serious and non-serious device-related events.

The primary outcome measure is hospital length of stay (LOS) defined as the number of days from hospital admission to the date the subject meets the medical elements of the GOLD Discharge Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Is over the age of 35 years
2. Has a history of COPD confirmed by physician diagnosis
3. Has been admitted to the hospital with a working diagnosis of acute exacerbation of COPD (AECOPD) defined as at least two of the following progressive symptoms: increased dyspnea, increased sputum volume and/or increased sputum purulence that is beyond normal day-to-day variation
4. Has a history of incomplete airway reversibility (e.g., patient not responding clinically to short-acting ß-agonists in the ED) associated with a diagnosis of COPD
5. Smoking history of at least 20 pack years
6. FEV1/FVC ratio of < 0.7 and impaired FEV1 (< 80% predicted for age, sex, race and height)
7. Is willing to participate in a 7 days post discharge (± 2 days) in-person follow-up visit and a telephone follow-up call 30 days (± 5 days) after hospital discharge
8. Is able to give written Informed Consent, or his/her legally authorized representative is available to give written Informed Consent

Exclusion Criteria:

1. Has a confirmed history of asthma (by pulmonary functions, response to ß-agonists and variable symptoms)
2. Has a history of lung cancer or Talc lung
3. Is admitted to the emergency care facility with a diagnosis of the following, confirmed on CXR, ventilation/perfusion scanning or computerized tomography (CT):

   * Pulmonary abscess;
   * Pneumonia (e.g., fever > 38.0° C, cough and new documented infiltrate)
   * Acute pulmonary embolism
   * Large pleural effusion and/or requiring thoracentesis; or
   * Pneumothorax
4. Is admitted to the emergency care facility with a working diagnosis of:

   * Acute coronary syndrome
   * Severe carotid artery disease (e.g., history of bruits, transient ischemic attack (TIA) or cerebrovascular accident (CVA); or
   * Stage IV heart failure according to the NYHA classification
5. Is admitted to the emergency care facility and/or hospital with a working diagnosis of:

   * Cystic Fibrosis; or
   * Tuberculosis
   * Pneumocystis carinii pneumonia (PCP) infection in the setting of HIV
6. Other severe cardiovascular acute diseases (such as uncontrolled hypertension, recent onset rapid atrial fibrillation and severe ventricular arrhythmias)
7. Is at risk of imminent respiratory collapse:

   * Lung Function: FEV1 < 25%
   * Rapid deterioration in respiratory status (sudden change in respiratory rate, decrease in oxygen saturation, change in consciousness, etc).
8. Has a condition in which collecting blood would be contraindicated or blood samples are unable to be obtained;
9. Has an abscess or other infection, lesion (including lymphadenopathy), surgical scar, congenital changes or broken skin at the treatment site on the neck;
10. Has confirmed severe sepsis or septic shock
11. Has a fever > 38.0° C
12. Has clinically significant changes in blood pressure or is receiving vasopressors to maintain blood pressure
13. Has an implanted electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, automated implantable cardioverter defibrillators (AICD), vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
14. Has a history of carotid endarterectomy or vascular neck surgery on the right side
15. Has implanted metal cervical spine hardware
16. Has a condition that would interfere with completing the self-assessment questionnaires
17. Is pregnant or breast feeding
18. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days
19. Belongs to a population or has any condition such that the investigator believes his or her ability to provide informed consent, comply with follow-up requirements or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be provided a study information sheet (informed consent form) to review. Those who are interested in participating will provide signed informed consent and then be screened for eligibility (inclusion/exclusion criteria). Subjects meeting the inclusion/exclusion criteria will be assigned a study ID number, randomized and enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rowe, M.D., Principal Investigator — University of Alberta
Locations (1):
- Edmonton Hospital, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- AlphaCore Active Device: AlphaCore device group will consist of subjects enrolled into the study with chronic obstructive pulmonary disease and receive an electrical stimulation to the vagus nerve to help open the subjects airways during the subjects stay in the hospital.
  AlphaCore Device: multiple stimulation treatments per day for duration of hospitalization
- AlphaCore Sham Device: AlphaCore Sham device group will consist of subjects enrolled into the study with chronic obstructive pulmonary disease, Sham device has no signal to the vagus nerve.
  AlphaCore ShamDevice: multiple stimulation treatments per day for duration of hospitalization
Period: Overall Study
Arm/Group | AlphaCore Active Device | AlphaCore Sham Device
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | AlphaCore Active Device | AlphaCore Sham Device | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66 [58 to 74] | 72 [65 to 79] | 69 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Length of Stay in the Hospital
Description: The primary outcome measure was hospital length of stay (LOS) defined as the number of days from hospital admission to the date the subject met the medical elements of the GOLD Discharge Criteria. (Global Initiative for Chronic Obstructive Lung Disease report, "Global Strategy for the Diagnosis, Management and Prevention of Chronic Obstructive Pulmonary Disease", Revised 2011)
Time Frame: Admission to hospital, 1 week in-person visit and a 30 day phone call follow-up visit from time of discharge from the hosptal
Population: Safety population
Measure: Mean (Full Range); unit: Days
Arm/Group | AlphaCore Active Device | AlphaCore Sham Device
Number analyzed (Participants) | 2 | 2
Days | 9 [7 to 11] | 5.5 [5 to 6]

ADVERSE EVENTS:
Time Frame: Admission to hospital, 1 week in-person visit and a 30 day phone call follow-up visit from time of discharge from the hosptal
Arm/Group | AlphaCore Active Device | AlphaCore Sham Device
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlphaCore Active Device (N=2) | AlphaCore Sham Device (N=2)
Non-ST elevation myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion/ Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Acute exacerbations of chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less